CLINICAL TRIAL: NCT01335672
Title: Survival After First Myocardial Infarction in Patients With and Without Chronic Obstructive Pulmonary Disease
Status: Completed | Type: Observational
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: British Medical Research Council (Other Government); University College, London (Other)
Responsible Party: Principal Investigator, Jennifer Quint, Senior Lecturer, London School of Hygiene and Tropical Medicine
Other Study IDs: 10-05; 086091/Z/08/Z (Other Grant/Funding Number: Wellcome)
Record Dates: First submitted 2011-04-12; First posted 2011-04-14 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Myocardial Infarction; Chronic Obstructive Pulmonary Disease
Keywords: Myocardial infarction; chronic obstructive pulmonary disease; General Practice Research Database; Myocardial Ischaemia National Audit Project; CALIBER
MeSH Terms: conditions — Myocardial Infarction; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- GPRD patients: All patients included in "up to standard" GPRD practices that agreed to the linkage with the MINAP database are included in this cohort.

SUMMARY:
An estimated three million people are affected by chronic obstructive pulmonary disease (COPD) in the UK, giving it a prevalence of 1.5% of the population in 2007/08. COPD accounts for approximately 30,000 deaths each year in the UK and is an important co-morbidity in those dying from other smoking related diseases, most commonly ischaemic heart disease and lung cancer. The National COPD audit showed a very high level of co-morbidity, the association with cardiovascular disease being particularly strong with 51% of patients with cardiovascular disease having been admitted for COPD within the preceding 24 months. Patients with COPD are at increased risk of myocardial infarction compared to the general population. Although this increase in cardiovascular risk exists, it is not clear is whether survival after myocardial infarction is different in patients with and without COPD and what factors contribute to this survival difference. Differences in survival may arise due to differences in prescribing certain drugs such as beta-blockers, differences in prevalence of risk factors (e.g. current smoking status) or increased COPD events such as exacerbations which themselves are associated with increased mortality.

The investigators primary aim is to investigate whether survival after first myocardial infarction is shorter in patients with COPD than those without COPD and to establish reasons for these differences in survival.

DETAILED DESCRIPTION:
This study is part of the CALIBER (Cardiovascular disease research using linked bespoke studies and electronic records) programme funded over 5 years from the NIHR and Wellcome Trust. The central theme of the CALIBER research is linkage of the Myocardial Ischaemia National Audit Project (MINAP) with primary care (GPRD) and other resources. The overarching aim of CALIBER is to better understand the aetiology and prognosis of specific coronary phenotypes across a range of causal domains, particularly where electronic records provide a contribution beyond traditional studies. CALIBER has received both Ethics approval (ref 09/H0810/16) and ECC approval (ref ECC 2-06(b)/2009 CALIBER dataset).

Objectives:

1. To investigate survival differences after first myocardial infarction in patients with and without COPD.
2. To investigate if these survival differences exist due to a) differences in prevalence of risk factors (e.g. smoking) b) differences in management after myocardial infarction (e.g. uptake of cardiac rehabilitation, prescription of beta-blockers) and c) COPD related events (e.g. exacerbations).

ELIGIBILITY:
Inclusion Criteria:

* Patients in GPRD practices which are deemed "up to standard" by GPRD criteria will be included if their practice agreed to be linked to the MINAP dataset.
* Age over 18.

Exclusion Criteria:

* Patients will be excluded after experiencing their first MI.
* Patients will be excluded if they do not fulfil one of the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is comprised of patients registered at those GPRD practices that agreed to the linkage with the MINAP database, and whose practices are "up to standard" according to GPRD criteria. Practices taking part in the GPRD are chosen to be representative of all UK practices, and 98% of people in the UK are registered with a GP. Therefore the GPRD should be a representative sample of the UK population
Sampling Method: Non-Probability Sample
Enrollment: 2100000 (Actual)
Dates: Start 2011-03; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Death after a first ST elevation or non ST elevation MI | Average time frame: patients in the GPRD are followed from registration until they experience the outcome, leave the practice, die, or 31st December 2009, whichever occurs first
  The primary outcome is death after a first ST elevation or non ST elevation MI. Death information will be based on data from one or more of the following: ONS death certificates; Hospital Episode Statistics; MINAP data; GPRD data.

SECONDARY OUTCOMES:
Number of patients with and without COPD prescribed a beta blocker after a MI | Average time frame: patients in the GPRD are followed from registration until they experience the outcome, leave the practice, die, or 31st December 2009, whichever occurs first
  Survival differences will be investigated with respect to a) differences in prevalence of risk factors (e.g. smoking) b) differences in management after myocardial infarction (e.g. uptake of cardiac rehabilitation, prescription of beta-blockers) and c) COPD related events (e.g. exacerbations).

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer K Quint, MRCP PhD, Principal Investigator — London School of Hygiene and Tropical Medicine; Harry Hemingway, FRCP, Study Director — University College, London
Locations (1):
- London School of Hygiene and Tropical Medicine, London, United Kingdom

REFERENCES:
- [Derived] Quint JK, Herrett E, Bhaskaran K, Timmis A, Hemingway H, Wedzicha JA, Smeeth L. Effect of beta blockers on mortality after myocardial infarction in adults with COPD: population based cohort study of UK electronic healthcare records. BMJ. 2013 Nov 22;347:f6650. doi: 10.1136/bmj.f6650. PMID 24270505